CLINICAL TRIAL: NCT01616914
Title: Delirium and Clinical Outcome
Brief Title: Subclinical Delirium and Clinical Outcome
Acronym: ZZH-2
Status: Completed | Type: Observational
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongheng Zhang, Jinhua central hospital, Jinhua Central Hospital
Other Study IDs: ZZH-2
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-06

CONDITIONS: Delirium
Keywords: delirium; outcome
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- delirium group: patients with delirium during ICU stay
- non-delirium group: patients without delirium during ICU stay

SUMMARY:
Delirium has been associated with clinical outcomes in critical care setting. However, its subclinical form has not been investigated. The investigators aimed to establish the association of subclinical delirium with outcome.

DETAILED DESCRIPTION:
Delirium has been associated with clinical outcome in critical care setting. This syndrome has been associated with longer length of stay in ICU and hospital, longer duration of mechanical ventilation and higher mortality rate. however, its subclinical form has not been investigated. The subclinical syndrome is defined by CAM-ICU, in which several features of delirium are fulfilled but the diagnostic criteria are not fulfilled. The investigators aimed to establish the association of subclinical delirium with outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients enter ICU
* GCS > 10
* RASS > -2

Exclusion Criteria:

* unable to cooperate
* coma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients enter ICU GCS > 10 RASS > -2 No dementia
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
mortality | during hospital stay(60 days)
  60 days after enrollment

SECONDARY OUTCOMES:
duration of mechanical ventilation | 60 days
length of stay in ICU and hospital | 60 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Zhongheng Zhang, MM, Study Chair — Jinhua Central Hospital
Locations (1):
- Jinhua central hospital, Jinhua, Zhejiang, China

REFERENCES:
- [Background] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509
- [Background] van den Boogaard M, Schoonhoven L, van der Hoeven JG, van Achterberg T, Pickkers P. Incidence and short-term consequences of delirium in critically ill patients: A prospective observational cohort study. Int J Nurs Stud. 2012 Jul;49(7):775-83. doi: 10.1016/j.ijnurstu.2011.11.016. Epub 2011 Dec 22. PMID 22197051
- [Background] Tomasi CD, Grandi C, Salluh J, Soares M, Giombelli VR, Cascaes S, Macedo RC, de Souza Constantino L, Biff D, Ritter C, Dal Pizzol F. Comparison of CAM-ICU and ICDSC for the detection of delirium in critically ill patients focusing on relevant clinical outcomes. J Crit Care. 2012 Apr;27(2):212-7. doi: 10.1016/j.jcrc.2011.05.015. Epub 2011 Jul 6. PMID 21737237